CLINICAL TRIAL: NCT02294604
Title: The Antiseptic Outcome of Traditional Hand Scrubbing Versus Hand Rubbing in Surgical Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Ka-Wai Tam, Director of Center for Evidence-Based Health Care, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 103HCP002
Record Dates: First submitted 2014-11-10; First posted 2014-11-19 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Hand Disinfection

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group R (Experimental): Waterless surgical hand rub formulation containing 61% ethyl alcochol, 1% chlorhexidine and moisturizers
  Interventions: Device: ethyl alcochol, chlorhexidine and moisturizers
- Group I (Active Comparator): Traditional scrub formation with 10 % povidone-iodine
  Interventions: Device: povidone-iodine
- Group C (Active Comparator): Traditional scrub formation with 4% chlorhexidine
  Interventions: Device: chlorhexidine

INTERVENTIONS:
Device: ethyl alcochol, chlorhexidine and moisturizers
  Other Names: Avagard
  Arms: Group R
Device: chlorhexidine
  Arms: Group C
Device: povidone-iodine
  Arms: Group I

SUMMARY:
Hand hygiene is the cornerstone of aseptic techniques to reduce surgical site infection. The traditional surgical antisepsis involves scrubbing the skin with povidone-iodine or chlorhexidine gluconate. Recently, a waterless surgical hand rub formulation containing 61% ethyl alcochol, 1% chlorhexidine and moisturizers was developed to provide a comparable antiseptic effect. The investigators perform a randomized controlled trial to compare the antiseptic effectiveness of the waterless hand rubbing, the classic surgical handwashing with povidone-iodine and chlorhexidine solutions.

DETAILED DESCRIPTION:
This single centre, randomized trial recruited surgical team members in Taipei Medical University-Shuang Ho Hospital at November 2014. 255 episodes of hand washing are enrolled. The participants are assigned equally to use either a waterless hand rub (Group R), or traditional scrub formation with 10 % povidone-iodine (Group I) and 4% chlorhexidine (Group C). Hand washing time, microorganisms on hands before and after scrubbing is recorded. The primary outcome is the colonies grown on bacterial culture plates and expressed as colony-forming units (CFU) on plates after hand washing. The secondary outcomes is hand microbial flora after surgery and duration of hand washing.

ELIGIBILITY:
Inclusion Criteria:

* Surgical staff members, both surgeons and scrub nurses

Exclusion Criteria:

* Participants were excluded if they were medical or nursing students
* Allergy to the experimental materials

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Wai Tam, MD, MS, Study Chair — Taipei Medical University Shuang Ho Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group R: Waterless surgical hand rub formulation containing 61% ethyl alcochol, 1% chlorhexidine and moisturizers
  ethyl alcochol, chlorhexidine and moisturizers
- Group I: Traditional scrub formation with 10 % povidone-iodine
  povidone-iodine
- Group C: Traditional scrub formation with 4% chlorhexidine
  chlorhexidine
Period: Overall Study
Arm/Group | Group R | Group I | Group C
Started | 80 | 80 | 80
Completed | 79 | 77 | 80
Not Completed | 1 | 3 | 0
Not completed — Did not provide samples for culture | 0 | 1 | 0
Not completed — Culture contamination | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group R | Group I | Group C | Total
Number analyzed (Participants) | 80 | 80 | 80 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 80 | 80 | 80 | 240
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants] — Gender was not assessed
  participants
    Unknown | 80 | 80 | 80 | 240
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 80 | 80 | 80 | 240
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 80 | 80 | 80 | 240

OUTCOME MEASURES:

1. Primary Outcome: Microorganisms on Hands Before Scrubbing
Description: The primary outcome is the colonies grown on bacterial culture plates and expressed as colony-forming units (CFU) on plates
Time Frame: 2 days after sampling
Measure: Mean (Standard Error); unit: colony forming unit
Arm/Group | Group R | Group I | Group C
Number analyzed (Participants) | 79 | 77 | 80
colony forming unit | 28.99 (3.98) | 38.64 (4.36) | 22.91 (3.63)

2. Secondary Outcome: Microorganisms on Hands After Scrubbing
Description: The secondary outcomes is the colonies grown on bacterial culture plates and expressed as colony-forming units (CFU) on plates
Time Frame: 2 days after sampling
Measure: Mean (Standard Error); unit: colony forming unit
Arm/Group | Group R | Group I | Group C
Number analyzed (Participants) | 79 | 77 | 80
colony forming unit | 1.38 (0.74) | 4.29 (1.25) | 0.48 (0.22)

3. Secondary Outcome: Microorganisms on Hands After Surgery
Description: The secondary outcomes is the colonies grown on bacterial culture plate
Time Frame: 2 days after sampling
Measure: Mean (Standard Error); unit: colony forming unit
Arm/Group | Group R | Group I | Group C
Number analyzed (Participants) | 79 | 77 | 80
colony forming unit | 4.7 (1.8) | 3.9 (1.6) | 4.1 (1.9)

4. Secondary Outcome: Duration of Hand Washing
Description: The secondary outcome is the duration of hand washing
Time Frame: Immediately
Measure: Mean (Standard Error); unit: Minute
Arm/Group | Group R | Group I | Group C
Number analyzed (Participants) | 79 | 77 | 80
Minute | 3.2 (0.2) | 3.64 (0.2) | 4.8 (0.8)

ADVERSE EVENTS:
Arm/Group | Group R | Group I | Group C
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/77 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/77 | 0/80
Other Adverse Events (participants affected / at risk) | 0/79 | 0/77 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No